CLINICAL TRIAL: NCT03143205
Title: Gene Expression Outcomes in Interventions for Substance Using HIV+ Minority Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23DA039800 (NIH); K23DA039800 (NIH)
Record Dates: First submitted 2017-05-02; First posted 2017-05-08 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-04

CONDITIONS: Human Immunodeficiency Virus Infection; Inflammation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AWARENESS for sexual minorities (Experimental): Group receives new CBT-based intervention
  Interventions: Behavioral: AWARENESS for Sexual Minorities
- Writing tasks (Active Comparator): Group receives writing-based sessions
  Interventions: Behavioral: Writing tasks

INTERVENTIONS:
Behavioral: AWARENESS for Sexual Minorities — 9 session, individually delivered, cognitive behavioral intervention focused on modifying sexual minority stress responses to reduce the impact of sexual minority stress experiences.
  Arms: AWARENESS for sexual minorities
Behavioral: Writing tasks — Writing sessions to explore daily activities.
  Arms: Writing tasks

SUMMARY:
This is a pilot study of a new 9-session individually delivered cognitive behavioral intervention targeting sexual minority stress. In this study, 40 HIV+ men sexual minority men will be recruited for the study then will be randomly assigned to either the new 9 session intervention or a writing task condition.

ELIGIBILITY:
Inclusion Criteria:

* Provide evidence or documentation of HIV positive status (e.g. a letter of diagnosis or medication bottles with matched photo ID)
* Be English speaking
* Be able to consent
* Sexual activity with a man in the 3 years prior to initial contact or identification as gay or bisexual
* Not currently be enrolled in formal substance abuse treatment
* Report at least one occasion of drinking 5 or more drinks or of using an illicit substance in the previous 3 months, but not meet criteria for a severe substance use disorder.

Exclusion Criteria:

* Presence of a severe substance use disorder
* Presence of current symptoms consistent with schizophrenia or bipolar disorder, which would indicate that an intervention targeting these symptoms would be more appropriate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant must self-identify as male at the time of screening into the study
Enrollment: 40 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Change in Gene expression | Baseline, ~9 weeks (at conclusion of intervention), 4 month follow-up
  Gene expression related to inflammation measured in blood

SECONDARY OUTCOMES:
Change in Substance Use | Baseline, ~9 weeks (at conclusion of intervention), 4 month follow-up
  Substance Use measured through Alcohol Smoking and Substance Involvement Screening Test (ASSIST)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Flentje A, Sunder G, Carrico AW, Asam K, Neilands TB, Lisha NE, Dilley J, Flowers E, Kober K, Aouizerat B. Differential gene expression in response to AWARENESS: A randomized controlled trial of an intersectional minority stress intervention. Health Psychol. 2025 Mar;44(3):291-296. doi: 10.1037/hea0001451. PMID 39992775